CLINICAL TRIAL: NCT07214714
Title: Hemodynamic and Cardiac Effects of Dexmedetomidine Versus Fentanyl by Intravenous Infusion as Adjuncts to General Anesthesia in Patients Undergoing Major Abdominal Cancer Surgeries.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nariman Khaled Abd Elmontalb Hamed, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dexmedetomidine versus fentany
Record Dates: First submitted 2025-10-05; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Abdominal Cancer Surgeries
MeSH Terms: interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group D (Active Comparator): Patients will receive Dexmedetomidineloading dose of 0.5 µg/kg over 10 minutes, followed by an infusion of 0.3-0.9 µg/kg/h.
  Interventions: Drug: Dexmedetomidine
- Group F (Active Comparator): Patients will receive Fentanyl loading dose of 1 µg/kg over 10 minutes, followed by an infusion of 0.5-1 µg/kg/h.
  Interventions: Drug: Fentanyl (IV)

INTERVENTIONS:
Drug: Fentanyl (IV) — Patients will receive Fentanyl loading dose of 1 µg/kg over 10 minutes, followed by an infusion of 0.5-1 µg/kg/h.
  Arms: Group F
Drug: Dexmedetomidine — Patients will receive Dexmedetomidine loading dose of 0.5 µg/kg over 10 minutes, followed by an infusion of 0.3-0.9 µg/kg/h.
  Arms: Group D

SUMMARY:
________________________________________

Background :

Major abdominal cancer surgery is among the most invasive procedures, often associated with extensive tissue damage, severe postoperative pain, and delayed recovery. Inadequate pain management can result in adverse physiological responses such as tachycardia, hypertension, prolonged immobility, and extended hospital stay. Moreover, poorly controlled pain may impair immune function and contribute to neuroendocrine, metabolic, gastrointestinal, and cardiopulmonary complications. Therefore, effective analgesia is essential to improve patient outcomes and recovery.

Multimodal analgesia has emerged as the gold standard for managing postoperative pain in major abdominal surgery. It integrates regional techniques (such as epidural or intrathecal analgesia), peripheral nerve blocks (e.g., transversus abdominis plane block), systemic opioids, and non-opioid agents including NSAIDs and acetaminophen. This approach minimizes surgical stress, maintains hemodynamic stability, and facilitates early ambulation and discharge.

Opioids, particularly fentanyl, are widely used as intrathecal adjuvants due to their rapid onset and favorable analgesic profile. However, selective alpha-2 adrenergic receptor agonists such as clonidine and dexmedetomidine are gaining attention for their sedative, analgesic, sympatholytic, and hemodynamic-stabilizing effects. Administered intrathecally, epidurally, or intravenously, they can enhance analgesia while reducing anesthetic requirements without causing profound sedation.

Conventional monitoring with heart rate and non-invasive blood pressure may overlook subtle variations in cardiac output. Electrical cardiometry (ICON®) provides continuous, non-invasive, beat-to-beat measurement of cardiac parameters and has been validated across different patient groups. Accordingly, the present study aims to compare intravenous dexmedetomidine and fentanyl as adjuvants to general anesthesia, focusing on their effects on hemodynamics and cardiac function in major abdominal cancer surgery using electrical cardiometry.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I- III, NYHA class I- II
* Patients subjected to elective major abdominal cancer surgeries.
* The enrolled age will be ≥ 18 years.

Exclusion Criteria:

* Unfit for surgery
* Patient refusal
* Body mass index>40 kg/m2
* ASA physical status IV-V, NYHA class III-IV.
* Chronic opioid consumption
* Contraindications to neuraxial block (coagulopathy, infection, or hematological disorders).
* Pregnant women
* Hypersensitivity to any of the used drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
cardiac output (CO) | 24 hour postoperative
  cardiac output (CO) measured using the non-invasive ICON® monitor